CLINICAL TRIAL: NCT07333911
Title: ORLINT & ORLEXT: New Orthosis for the Lateral Knee Ligaments
Brief Title: ORLINT & ORLEXT: Orthosis for Knee
Acronym: ORLINT&ORLEXT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Rocío Llamas-Ramos, Principal Investigator, University of Salamanca
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Device Feasibility
Other Study IDs: ORLINT&ORLEXT2026; University of Salamanca (Other Grant/Funding Number: University of Salamanca)
Record Dates: First submitted 2025-12-08; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Knee Brace; Knee

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orlint-Orlext orthosis group (Experimental): Participants must wear the new knee orthosis during assessments and in their daily lives for at least one month, which is the duration of the study.
  Interventions: Device: Orlint-Orlext orthosis device
- Conventional orthesis group (Active Comparator): Participants must wear the conventional knee orthosis (a without orthosis) during assessments and in their daily lives, before wear the new one.
  Interventions: Device: Conventional orthosis device

INTERVENTIONS:
Device: Orlint-Orlext orthosis device — Participants must wear the new knee orthosis during assessments and in their daily lives for at least one month, which is the duration of the study.
  Arms: Orlint-Orlext orthosis group
Device: Conventional orthosis device — Participants must wear the conventional knee orthosis and without orthosis, during assessments and before wearing the new one
  Arms: Conventional orthesis group

SUMMARY:
The goal of this experimental study is to test the feasibility and validity of a new orthosis in patients with lateral ligament knee lesions of both sexes and older than 18 years old. The main question it aims to answer is:

Is the new orthosis a support for knee stability?? Does the new orthosis improve knee function and patients' quality of life??

The control group will be the subjects themselves when wearing their conventional knee orthosis or without it.

Participants must wear the new knee orthosis for at least one month to assess the effectiveness of the orthosis and evaluate any changes that have occurred in the knee joint and muscles.

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic knee injuries
* patients who have already been prescribed an orthosis
* patients older than 18 years old

Exclusion Criteria:

* inability to stand actively and stably
* inability to walk unaided

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Device feasibility | Baseline and up to 4 weeks
  Device feasibility will be assessed through participants' awareness of the device, as an indicator of its accessibility, visibility, and potential for effective implementation within the target population. A self-diary will be requested

SECONDARY OUTCOMES:
Knee function with virtual reality | Baseline and up to 4 weeks
  Knee function will be assessed using a virtual reality programme that requires movement of the lower limb to assess knee stability, with and without orthosis. The assessment will be using a Borg scale (range of effort that the individual perceives when exercising). From 0 points (minimum effort) to 10 points (maximum effort).
Range of motion with a Gyko device | Baseline and up to 4 weeks
  The range of motion of the knee joint will be measured using the Gyko device with and without the new orthosis. It will be measured in degrees (0-120º)
Footprint with a pressure platform | Baseline and up to 4 weeks
  The distribution of static and dynamic load will be assessed with and without orthosis, using a pressure platform, as well as static balance with eyes open and closed and dynamic balance. The meausure will be the percentaje of support from the sole of the foot.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Salamanca, Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No